CLINICAL TRIAL: NCT03338777
Title: Phase 1 Suicide Plus Immune Gene Therapy for Advanced Melanoma
Brief Title: Suicide Plus Immune Gene Therapy for Advanced Melanoma
Acronym: IGTM-101
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Failure to achieve primary objective
Sponsor: Hospital Italiano de Buenos Aires (Other)
Collaborators: Instituto de Oncología Ángel H. Roffo (Other); National Agency for Scientific and Technological Promotion, Argentina (Other); National Council of Scientific and Technical Research, Argentina (Other Government); University of Buenos Aires (Other)
Responsible Party: Principal Investigator, Simonovich Ventura, MD, Medical Doctor, Hospital Italiano de Buenos Aires
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2082
Record Dates: First submitted 2017-10-10; First posted 2017-11-09 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Melanoma
Keywords: melanoma; lipoplexes; plasmid; herpes simplex thymidine kinase; interleukin-2; granulocyte-macrophage colony-stimulating factor; tumor vaccine; suicide gene
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Intervention Model Description: Suicide plus immunogene therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Suicide plus immunogene therapy (Experimental): Intra and peritumoral infiltrates with multiple injections of lipoplexes carrying the HSVtk suicide gene co-administered with GCV and subcutaneous vaccine produced with formolized allogeneic tumor extracts and lipoplexes carrying hIL-2 and hGM-CSF genes.
  Interventions: Biological: Suicide plus immunogene therapy

INTERVENTIONS:
Biological: Suicide plus immunogene therapy — 1. Intra and peritumoral infiltrates with multiple injections of 0.1 ml/cm2 or 0.2 ml/cm3 of lipoplexes bearing the HSVtk suicide gene (1: 1; 1 mg/ml, according to tumor size), co-administered with GCV (12.5 mg/ml). Patients start with a minimum of 0.5 ml and at the 3rd week, the maximum dose is scaled according to the tumor size up to 2 ml maximum.
  2. Treated simultaneously with a subcutaneous vaccine produced with:
     * Formolized allogeneic tumor extracts and,
     * Lipoplexes carrying hIL-2 and hGM-CSF genes (0.5 mg each).

SUMMARY:
Safety evaluation of combined immunogene therapy in patients with advanced melanoma.

DETAILED DESCRIPTION:
This phase I clinical protocol is proposed to evaluate the safety of combined immunotherapy genetics in humans.

This treatment combines the high local cytotoxicity of the suicide gene system (HSV thymidine kinase: HSVt k) / prodrug (ganciclovir: GCV) with the immunostimulation of interleukin2 (hIL2) and immunoamplification of granulocyte and macrophage colony stimulating factor (hGMCSF) in the presence of tumor antigens.

The proposed scheme consists in the periodic intra / peritumoral application of plasmid DNA complexes: cationic lipid (lipoplexes) containing the HSVtk gene, co-administered with the prodrug GCV, and subcutaneous injections of a vaccine (LGvax) produced with formolized extracts of allogeneic melanoma combined with lipoplexes carrying the hIL2 and hGMCSF genes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically and / or cytologically confirmed melanoma.
* Patients progressed or are intolerant to conventional systemic treatments.
* Patients that are not candidates for surgery under oncologic criteria (complete resection).
* Performance status (ECOG) 0 or 1.
* Patients with life expectancy greater than 6 months.
* Patients with at least one accessible target lesion for gene inoculation (superficial localizations of the primary tumor, satelitosis, subcutaneous or accessible lymph node metastasis).
* Patients with measurable disease (according to RECIST 1.1 criteria, irrespective of the target lesion chosen for suicide gene inoculation)
* Patients with signed informed consent.

Exclusion Criteria:

* Patients with uncontrolled cardiovascular disease
* Patients with uncontrolled respiratory disease.
* Patients with uncontrolled immune disease.
* Patients with glucocorticoids or immunosuppressive drugs or agents with immunomodulatory activity (except non-steroidal anti-inflammatory agents) up to 2 weeks before treatment.
* Patients performing other experimental therapies.
* Patients who are pregnant or breastfeeding.
* Patients undergoing concurrent chemotherapy or radiation therapy.
* Uncontrolled diabetes.
* Patients with active diagnosis of other malignant neoplasms.
* HIV-positive patients.
* Uncontrolled thyroid abnormality.
* Patients with significant medical morbidity.
* Patients with a history of allergic reactions to chemicals or similar to those used in this study.
* Metastasis in the central nervous system.
* Laboratory eligibility criteria excluded:

  * Hemoglobin: <8 g / dL, leukocytes: <3,000 / mm3, platelets: <100,000 / mm3, neutrophils: <1000 / mm3, hematocrit: <25%. bilirubin> 2.0 mg / dL, GOT or GPT: 2.5 times> than normal upper institutional limit (ULN), alkaline phosphatase: 2 times> ULN, creatinine> 2.0 mg / dL, creatinine clearence : <60 ml / min / 1.73 m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Safety reported as the number of treatment-related adverse events as assessed by CTCAE v4.03 | 1 year
  Number of participants with treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03 (https://evs.nci.nih.gov/ftp1/CTCAE/CTCAE_4.03_2010-06-14_QuickReference_5x7.pdf).

CONTACTS AND LOCATIONS:
Overall Officials: Ventura Simonovich, MD, Principal Investigator — Hospital Italiano
Locations (1):
- Hospital Italiano, Ciudad Autónoma de Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No